CLINICAL TRIAL: NCT03920605
Title: Study on Optimized Treatment of Peginterferon Alfa 2a or 2b in Anti-virus Treatment Experienced Patients With Hepatitis b Virus Related Liver Fibrosis
Brief Title: Optimized Treatment of Peginterferon Alfa 2a/2b in Treatment Experienced Patients With HBV Related Liver Fibrosis
Acronym: HBV
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Liang Peng, Professor, Third Affiliated Hospital, Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PL5
Record Dates: First submitted 2019-04-16; First posted 2019-04-19 (Actual); Last update posted 2019-05-22 (Actual); Status verified 2019-05

CONDITIONS: Hepatitis B; Liver Fibrosis
Keywords: hepatitis b virus; peginterferon alfa; liver fibrosis
MeSH Terms: conditions — Hepatitis B; Liver Cirrhosis | interventions — Tenofovir; peginterferon alfa-2a; peginterferon alfa-2b

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Peginterferon alfa group (Active Comparator): 50 patients would receive treatment of subcutaneous injection of peginterferon alfa 2a 180 μg or peginterferon alfa 2b 80μg once per week from baseline to 48 weeks. Then they would receive treatment of oral tenofovir disoproxil fumarate (TDF) 300 mg once per day from 49 to 144 weeks.
  Interventions: Drug: Peginterferon Alfa-2a; Drug: Peginterferon Alfa-2b
- Combination group (Active Comparator): 50 patients would receive treatment of subcutaneous injection of peginterferon alfa 2a 180 μg or peginterferon alfa 2b 80μg once per week and meanwhile oral tenofovir disoproxil fumarate (TDF) 300 mg once per day from baseline to 48 weeks. Then they would receive treatment of oral TDF 300 mg once per day from 49 to 144 weeks.
  Interventions: Drug: Tenofovir Disoproxil Fumarate; Drug: Peginterferon Alfa-2a; Drug: Peginterferon Alfa-2b

INTERVENTIONS:
Drug: Tenofovir Disoproxil Fumarate — Patients would receive oral Tenofovir Disoproxil Fumarate 300mg once per day.
  Other Names: Viread
  Arms: Combination group
Drug: Peginterferon Alfa-2a — Patients would receive subcutaneous injection of Peginterferon Alfa-2a 180 μg once per week.
  Other Names: Pegasys
Drug: Peginterferon Alfa-2b — Patients would receive subcutaneous injection of Peginterferon Alfa-2b 80 μg once per week.
  Other Names: Pegintron

SUMMARY:
Compared to nucleoside/nucleotide analogues, peginterferon alfa 2a/2b may has more therapeutic efficacy in hepatitis B surface antigen or e antigen seroconversion and anti-tumor occurrence in chronic hepatitis b patients. We design this study to investigate treatment of peginterferon alfa 2a/2b in anti-virus treatment experienced patients with HBV related liver fibrosis.

DETAILED DESCRIPTION:
Compared to nucleoside/nucleotide analogues, peginterferon alfa 2a/2b may has more therapeutic efficacy in hepatitis B surface antigen or e antigen seroconversion and anti-tumor occurrence in chronic hepatitis b patients. But there still lacks of studies on peginterferon alfa 2a or 2b treatment in patients with HBV related liver fibrosis. We design this study to investigate optimized treatment of peginterferon alfa 2a/2b, comparing to nucleoside/nucleotide analogues, in anti-virus treatment experienced patients with HBV related liver fibrosis.

ELIGIBILITY:
Inclusion Criteria:

1. Positive hepatitis b surface antigen or hepatitis b virus DNA > 0.5 year;
2. Age from 18 to 55 years old;
3. Fibrosis lever of F1 to F3 from liver biopsy; if liver biopsy unreachable, fibrosis lever of 7 to 14 kpa from fibroscan;
4. Portal vein diameter ≤ 12 mm from liver ultrasound;
5. Receiving treatment of nucleoside/nucleotide analogues at the past one year;
6. Normal liver function;
7. Undetectable hepatitis b virus DNA.

Exclusion Criteria:

1. Decompensated cirrhosis, hepatocellular carcinoma or other malignancy;
2. Pregnancy or lactation;
3. Other active liver diseases；
4. Human immunodeficiency virus infection or congenital immune deficiency diseases;
5. Severe diabetes, autoimmune diseases;
6. Other important organ dysfunctions;
7. Patients can not follow-up;
8. Investigator considering inappropriate.

Ages: 15 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-02-01 (Actual); Primary Completion 2021-10-30 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Change of level of liver fibrosis after anti-virus treatment | 48 week, 144 week
  Liver biopsy or fibroscan would be accessed to know the change of level of liver fibrosis at 48 and 144 weeks after anti-virus treatment.

SECONDARY OUTCOMES:
Ratio of patients with undetectable hepatitis b virus DNA after anti-virus treatment | 24 week, 48 week, 72 week, 96 week, 120 week,144 week
  Hepatitis b virus DNA would be tested to know the ratio of patients with undetectable hepatitis b virus DNA at 6 time points after anti-virus treatment.
Ratio of patients with hepatitis b e antigen seroconversion after anti-virus treatment | 24 week, 48 week, 72 week, 96 week, 120 week,144 week
  Hepatitis b e antigen and hepatitis b e antibody would be tested to know the ratio of patients with negative hepatitis B e antigen and positive hepatitis B e antibody at 6 time points after anti-virus treatment.
Ratio of patients with hepatitis b surface antigen seroconversion after anti-virus treatment | 24 week, 48 week, 72 week, 96 week, 120 week,144 week
  Hepatitis b surface antigen and hepatitis b surface antibody would be tested to know the ratio of patients with negative hepatitis B surface antigen and positive hepatitis B surface antibody at 6 time points after anti-virus treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Liang Peng, Doctor, Principal Investigator — Third Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- Third Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China